CLINICAL TRIAL: NCT05919381
Title: A Randomized, Double-blind, Parallel Controlled Phase III Study of Gentuximab Injection Combined With Paclitaxel Injection Versus Placebo Combined With Paclitaxel Injection for Advanced Gastric or Gastroesophageal Junction Adenocarcinoma.
Brief Title: Gentuximab Combined With Paclitaxel Compared With Placebo Combined With Paclitaxel for Gastric Adenocarcinoma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gensci043-GC-III01
Record Dates: First submitted 2023-03-22; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2022-12

CONDITIONS: Adenocarcinoma of Stomach
Keywords: Adenocarcinoma of stomach or gastroesophageal junction.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentuximab Injection (Experimental): Gentuximab Injection 8 mg/kg, D1, 15 intravenous drip, combined with Paclitaxel Injection 80 mg/m2/time, D1, 8, 15 intravenous drip, a cycle every 28 days.
  Interventions: Drug: Gentuximab Injection; Drug: Gentuximab Injection Placebo
- Gentuximab Injection Placebo (Placebo Comparator): Gentuximab Injection Placebo 8 mg/kg, D1, 15 intravenous drip, combined with Paclitaxel Injection 80 mg/m2/time, D1, 8, 15 intravenous drip, a cycle every 28 days.
  Interventions: Drug: Gentuximab Injection; Drug: Gentuximab Injection Placebo

INTERVENTIONS:
Drug: Gentuximab Injection — Gentuximab Injection 8 mg/kg, D1, 15 intravenous drip, a cycle every 28 days.
Drug: Gentuximab Injection Placebo — Gentuximab Injection Placebo 8 mg/kg, D1, 15 intravenous drip, a cycle every 28 days.

SUMMARY:
To evaluate the efficacy and safety of the combination of Gentuximab Injection and Paclitaxel Injection in patients with advanced gastric or gastroesophageal junction adenocarcinoma after first-line treatment failure compared with Placebo and Paclitaxel Injection.

DETAILED DESCRIPTION:
It was planned to enroll 752 subjects, grouped according to a 1:1 ratio, with 376 cases each in the experimental group and the control group.

Screening period:

Screening period assessments were performed within 28 days prior to randomization. Patients are screened after signing the informed consent form (ICF), complete relevant laboratory tests and imaging evaluations (including physical examination, vital signs, height, weight, ECOG score, laboratory tests, 12-lead ECG, echocardiography, chest, abdomen, pelvic contrast/contrast CT and head enhancement MRI, whole body bone scan, etc.), and subjects who meet the inclusion criteria and do not meet the exclusion criteria can be enrolled.

Treatment period:

All eligible participants were randomly assigned to the following two groups in a 1:1 ratio based on stratified factors (time to randomization < 6 months or ≥ months from the start of first-line therapy):

1. Test group: Gentuximab injection 8 mg/kg, D1, 15 intravenous drip, combined with Paclitaxel injection 80 mg/m2/time, D1, 8, 15 intravenous drip, every 28 days.
2. Control group: placebo 8 mg/kg, D1, 15 intravenous drip, combined with paclitaxel injection 80 mg/m2/time, D1, 8, 15 intravenous drip, every 28 days.

Efficacy and quality of life scores were assessed every 8 weeks ± 7 days according to RECIST 1.1, including chest, abdomen, and pelvis. The safety profile of subjects throughout treatment was evaluated according to NCI-CTCAE V 5.0 criteria, including vital signs, physical examination, ECOG score, laboratory tests, 12-lead ECG, echocardiogram, adverse events, serious adverse events, etc.

Follow-up periods:

Follow-up periods include safety and survival follow-up, immediately after the last study drug is completed.

Safety follow-up: All subjects had a safety follow-up within 28±5 days after the last dose or before starting new antitumor therapy (except for subjects withdrawing informed consent, voluntary withdrawal, loss to follow-up, death, etc.), and performed vital signs, physical examination, weight, ECG score, 12-lead ECG, laboratory tests, etc. (see Table 1.3-1 for details), and recorded concomitant medication and adverse events. If safe follow-up is less than 14 days from the end of treatment (EOT) visit, EOT visit can be an alternative to safe follow-up without repeating.

Survival follow-up: For any subject who ends treatment due to non-disease progression (and does not take other antitumor therapy), it is still necessary to return to the hospital every 8 weeks ± 7 days according to the original tumor evaluation plan for tumor imaging evaluation and life scale evaluation until disease progression, start of new antitumor therapy, withdrawal of informed consent, voluntary withdrawal, loss to follow-up, death, etc. For participants whose disease has progressed or who have started new antineoplastic therapy, survival follow-up is recorded every 8 weeks ±7 days from the time of notification of disease progression or initiation of new antineoplastic therapy (telephone follow-up) and details of subsequent treatment regimens (antineoplastic therapy received after the end of the study drug) until death, loss to follow-up, or the end of the study (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* 18~75 years old (including boundary value), male and female.
* Patients with advanced gastric cancer or gastroesophageal junction adenocarcinoma diagnosed by histology have developed disease after receiving first-line treatment containing platinum and fluorouracil for at least one cycle.
* It is necessary to make sure that the Her-2 expression status is negative or Her-2 positive and fails to be treated with anti-Her-2 targeted drugs.
* There is at least one measurable focus according to the RECIST 1.1 evaluation criteria for the efficacy of solid tumors.
* The physical condition score of the Eastern Cancer Cooperation Group (ECOG) was 0 or 1.
* The expected life is at least 3 months.
* Weight ≥ 40 kg, or BMI ≥ 17.

Exclusion Criteria:

•• Have received any systemic treatment targeting VEGF or VEGFR signal pathway.

* Have received systemic treatment of paclitaxel, docetaxel and paclitaxel for injection (albumin binding type).
* Those who are allergic to antibody-like recombinant protein drugs, paclitaxel and its excipients.
* Have received chemotherapy, radiotherapy, molecular targeted therapy, immunotherapy and other systemic anti-tumor treatment within 4 weeks before the first administration or within 5 half-lives of the drug.
* Have undergone major surgery within 4 weeks before the first administration.
* Thromboembolism occurred within 6 months before screening.
* Be receiving anticoagulant treatment with warfarin or similar preparations.
* Severe hemorrhagic disease, vasculitis or gastrointestinal bleeding within 3 months before screening.
* There was a history of gastrointestinal perforation and/or fistula, a history of intestinal obstruction, and a history of inflammatory bowel disease within 6 months before screening.
* Have a serious history of cardiovascular disease.
* Symptomatic central nervous system metastasis.
* Other malignant tumors confirmed and/or requiring treatment in the past 3 years.
* Be suffering from infectious diseases.
* Have an immune system disease or mental illness that requires treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
OS | 36 months.
  From date of randomization until the date of first documented death from any cause,assessed up to 36 months.

SECONDARY OUTCOMES:
PFS | 36 months.
  From date of randomization until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 36 months.
TTF ORR DCR DOR | 36 months. 36 months. 36 months. 36 months.
  TTF:From date of randomization until the date of first documented progression or date of death from any cause or date of discontinuation of treatment due to AE, refusal of treatment, or other reasons (excluding due to good outcomes) ,whichever came first, assessed up to 36 months.
  ORR: Overall optimal response was the proportion of participants with CR or PR, assessed up to 36 months.
  DCR: From date of first assessment is CR or PR to the first assessment is PD or death from any cause, whichever came first, assessed up to 36 months.
  DOR: Overall optimal response was the proportion of participants with CR or PR or SD, assessed up to 36 months.

OTHER OUTCOMES:
Change form baseline in EORTC QLQ-C30. | 36 months.
  Change in EORTC QLQ-C30 until the date of first documented progression , assessed up to 36 months.
Change form baseline in EQ-5D-3L. | 36 months.
  Change in EQ-5D-3L until the date of first documented progression , assessed up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai Dongfang Hospital
Locations (1):
- Shanghai Dongfang Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Drugs belong to the sponsor before they are put into clinical trials and the site is only a contract research organization; It is an industry practice that intellectual property rights belong to the sponsor.